CLINICAL TRIAL: NCT03780478
Title: Evaluation of a Preoperative Nerve Block in Pain Scores Following Rhinoplasty/Septoplasty
Brief Title: Preoperative Nerve Block for Rhinoplasty/Septoplasty
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Amit Kochhar, Clinical Assistant Professor of Otolaryngology -Head & Neck Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rhinoplasty Nerve Block Study
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Nasal Fracture; Deviated Nasal Septum
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Intervention Model Description: rhinoplasty/septoplasty patients will be identified by Dr. Kochhar (PI). Patients' informed consent for participation in this study will be obtained and they will subsequently be enrolled. Participants will be randomized into two arms: experimental vs. placebo.
  Study arms:
  1. Experimental: SPG block with local anesthetic per normal methods of nerve block.
  2. Placebo: Injection of saline
Who Masked: Participant
Masking Description: After giving consent to participate in study, patients enrolled in study will be randomly assigned to either the experimental vs. normal standard of care. Patients and members of care team will be unaware as to which group they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SPG Block (Experimental): Sphenopalatine ganglion block
  Interventions: Drug: Nerve block
- Placebo Control (Placebo Comparator): Saline injection
  Interventions: Drug: Placebo Saline Injection

INTERVENTIONS:
Drug: Nerve block — 0.25% bupivacaine with epinephrine (1:100k), with total volume of 2mL
  Arms: SPG Block
Drug: Placebo Saline Injection — Saline injection, total volume 2ml
  Arms: Placebo Control

SUMMARY:
Addiction is an inherent risk when prescribing opiates for pain relief, and methods to reduce its use or amount prescribed can help mitigate this risk for addiction. Patients undergoing rhinoplasty are often prescribed a short course of opiates during the acute post surgical phase. Studies have shown intraoperative sphenopalatine ganglion (SPG) nerve block in endoscopic sinus surgery can reduce post operative narcotic use. The purpose of this study is to determine if use of SPG block can be used to reduce narcotic use in the acute post operative phase of rhinoplasty/septoplasty.

DETAILED DESCRIPTION:
With the current opioid epidemic, more than 40,000 deaths can be attributed to prescription and illicit opioid use per year. There is inherent risk for patients to develop addiction when prescribing opiates for pain relief, and methods to reduce its use or the amount prescribed can help mitigate this risk.

Surgery is one of the leading causes for prescribing narcotics to control pain. Patients undergoing rhinoplasty are often prescribed a short course of opiates during the acute post surgical phase. Intraoperative sphenopalatine ganglion (SPG) block has been successfully and safely used in endoscopic sinus surgery, and has been shown to decrease narcotic use and inpatient hospital stay time.

The investigators are interested in determining if use of SPG block may offer an improved strategy to reducing the use of narcotics for post rhinoplasty/septoplasty pain relief. The investigators hypothesize that SPG block will reduce the amount of post operative opiates required for pain control.

The study population will include patients undergoing rhinoplasty/septoplasty at Keck Medical Center of USC who are able to provide consent. The study will include two arms: SPG block (experimental) and placebo saline injection (control). Patients' post operative pain scale and narcotic use will be recorded until first follow-up visit (2 weeks). Patient demographics, surgical indication, and intraoperative analgesia will be recorded. T-tests will be conducted between patient groups. ANOVA will be used to analyze other factors that may be associated with decreased narcotic use.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient requiring rhinoplasty/septoplasty and able to provide consent.
2. Must be willing to participate.
3. Must be able to complete consent in English or Spanish.

Exclusion Criteria:

1. History of opioid substance abuse disorder.
2. <18 years old
3. Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Post op Narcotic Use | 7 days
  Amount of narcotic use in post operative phase will be recorded until follow up visit
Post op Numerical pain scale | 7 days
  Pain scale will be recorded daily until follow up visit. Pain scale is defined as 0-10, where 0 is no pain, and 10 is worst pain ever experienced. Pain score will be obtained daily, and experimental arm will be compared with control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Kochhar, MD, Principal Investigator — USC Keck Medical Center
Locations (1):
- Keck Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Qudah M. Endoscopic sphenopalatine ganglion blockade efficacy in pain control after endoscopic sinus surgery. Int Forum Allergy Rhinol. 2016 Mar;6(3):334-8. doi: 10.1002/alr.21644. Epub 2015 Sep 15. PMID 26370724
- [Background] DeMaria S Jr, Govindaraj S, Chinosorvatana N, Kang S, Levine AI. Bilateral sphenopalatine ganglion blockade improves postoperative analgesia after endoscopic sinus surgery. Am J Rhinol Allergy. 2012 Jan-Feb;26(1):e23-7. doi: 10.2500/ajra.2012.26.3709. PMID 22391074
- [Background] Kesimci E, Ozturk L, Bercin S, Kiris M, Eldem A, Kanbak O. Role of sphenopalatine ganglion block for postoperative analgesia after functional endoscopic sinus surgery. Eur Arch Otorhinolaryngol. 2012 Jan;269(1):165-9. doi: 10.1007/s00405-011-1702-z. Epub 2011 Jul 8. PMID 21739090
- [Background] Patel S, Sturm A, Bobian M, Svider PF, Zuliani G, Kridel R. Opioid Use by Patients After Rhinoplasty. JAMA Facial Plast Surg. 2018 Jan 1;20(1):24-30. doi: 10.1001/jamafacial.2017.1034. PMID 29121158
- See also: 6) National Institue on Drug Abuse. Overdose Death Rates. NIDA. — https://www.drugabuse.gov/related-topics/trends-statistics/overdose-death-rates
- See also: Role of Intraoperative Endoscopic Sphenopalatine Ganglion Block in Sinonasal Surgery — https://scialert.net/abstract/?doi=jms.2007.1297.1303